CLINICAL TRIAL: NCT00125853
Title: A Trial to Compare the Effects of Nebivolol Versus Atenolol on Various Cardiovascular Measurements Including Insulin Sensitivity
Brief Title: The Effect of Nebivolol on Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Foundation for Circulatory Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NPSW02
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Hypertension
Keywords: blood pressure; insulin sensitivity; beta blockers; randomised double blind crossover trial
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — Nebivolol; Atenolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atenolol 25mg daily (Experimental): atenolol 25mg daily
  Interventions: Drug: Atenolol
- nebivolol 2.5mg daily (Active Comparator): nebivolol 2.5mg daily
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 2.5mg daily
  Arms: nebivolol 2.5mg daily
Drug: Atenolol — Atenolol 25mg daily
  Arms: atenolol 25mg daily

SUMMARY:
The purpose of this study is to conduct a randomised trial to compare the insulin sensitivity, 24 hour blood pressure profile, and tolerability of nebivolol plus a thiazide-like diuretic versus atenolol plus a thiazide-like diuretic.

DETAILED DESCRIPTION:
Retrospective studies of treated hypertensive cohorts have strongly implicated beta blocker therapy as increasing the risk of developing new-onset diabetes. This has led to the latest British Hypertension Society guidelines advising caution when using beta blockers particularly in combination with thiazide-like diuretics. However the National Institute of Clinical Excellence recommends beta-blocker + thiazide combinations as the treatment of choice in patients who are not at increased risk of developing diabetes. Nebivolol is a newer class of beta blocker. Some studies in diabetic hypertensive patients have suggested that nebivolol does not impair insulin sensitivity. The aim of this study is to compare the effect on insulin sensitivity of nebivolol versus atenolol, both in combination with a thiazide-like diuretic, in a group of non-diabetic hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 or above
* Blood pressure that meets any of the three following criteria:
* BP should be <140/85 mmHg on a maximum of two anti-hypertensive drugs

Exclusion Criteria:

* contraindications to beta-blockade
* contraindications to thiazide use
* if there was a history of asthma, diabetes, heart failure, bradycardia, atrial fibrillation, AV conduction disturbances
* concurrent treatment with verapamil & dilitiazem
* childbearing women
* compelling indication for treatment with a beta blocker
* any condition that will interfere with the treatment or the patient's ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R Poulter, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Paddington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- First is Atenolol Followed by Nebivolol (AN): Atenolol 25mg daily for 8 weeks, followed by a 4-week wash-out period, then nebivolol 2.5 mg daily for 8 weeks
- First is Nebivolol Followed by Atenolol (NA): Nebivolol 2.5mg daily for 8 weeks, followed by a 4-week wash-out period, then atenolol 25 mg daily for 8 weeks
Period: Wash-out (4 Weeks)
Arm/Group | First is Atenolol Followed by Nebivolol (AN) | First is Nebivolol Followed by Atenolol (NA)
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: First Intervention (8 Weeks)
Arm/Group | First is Atenolol Followed by Nebivolol (AN) | First is Nebivolol Followed by Atenolol (NA)
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Wash-out (4 Weeks)
Arm/Group | First is Atenolol Followed by Nebivolol (AN) | First is Nebivolol Followed by Atenolol (NA)
Started | 27 | 27
Completed | 24 | 20
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7
Period: Second Intervention (8 Weeks)
Arm/Group | First is Atenolol Followed by Nebivolol (AN) | First is Nebivolol Followed by Atenolol (NA)
Started | 24 | 20
Completed | 24 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Crossover study design all participants will receive both treatments
Arm/Group | All Participants
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 25
BMI [Mean (Standard Deviation); unit: kg/m^2] — kg/m2
  kg/m^2 | 27.2 (6.7)
Current Smoker [Count of Participants; unit: Participants] | 14
Ex-smoker [Count of Participants; unit: Participants] | 14
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 129.4 (13.2)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 81.3 (9.0)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 71.1 (8.9)
HBa1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.7 (0.7)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Index (ISI)
Description: Patients were asked to fast for a minimum of 12 hours prior to each oral glucose tolerance test (OGTT). Venous blood was withdrawn for insulin and glucose analysis, 15 minutes and immediately prior to, and 30, 60, 90 and 120 minutes following an oral glucose load. For each OGTT, the Insulin Sensitivity Index (ISI) was calculated using the standard method for oral glucose tolerance testing.
  For each OGTT, the Insulin Sensitivity Index (ISI) was calculated using the standard method for oral glucose tolerance testing.
Time Frame: Baseline, 15, 30, 60, 90, 120m following oral glucose load, at baseline and at the end of each phase(8 weeks treatment
Population: Patients with mild-to-moderate essential hypertension, aged 18 years or above, with blood pressure controlled to <140/85 mmHg on a maximum of two antihypertensive drugs, were recruited from the Peart-Rose Hypertension clinic at St Mary's Hospital in West London and from local general practices.
Measure: Mean (Inter-Quartile Range); unit: factor
Groups:
- Atenolol: Participants received Atenolol 25mg daily for 8 weeks
- Nebivolol: Participants received Nebivolol 2.5mg daily for 8 weeks
Arm/Group | Atenolol | Nebivolol
Number analyzed (Participants) | 44 | 44
factor
  Before | 82.36 [50.8 to 116.9] | 80.70 [52.6 to 114.7]
  After | 75.47 [50.6 to 144.9] | 81.54 [50.9 to 114.9]
Statistical Analysis 1: Comparison: Atenolol vs Nebivolol; Comparing treatment effects on ISI; Test type: Other — Linear Mixed effect Modelling, adjusted for baseline values and period effect Difference of LSMeans treatment effect (SE) = 0.05 (0.09); p = 0.60, Linear Mixed effect Modelling, adjusted

2. Secondary Outcome: 24 Hour Systolic Blood Pressure
Description: The 24-h Ambulatory Blood Pressure Monitoring (ABPM) was recorded at the beginning and end of each beta-blocker treatment period. BP was automatically recorded for 24 h at 30 min intervals. The time periods from 0700h to 2200h and from 2200h to 0700h were defined as daytime and night-time, respectively.
Time Frame: Before and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Atenolol | Nebivolol
Number analyzed (Participants) | 44 | 44
mmHg
  SBP before | 128.4 (9.7) | 130.4 (9.5)
  SBP after | 117.2 (9.2) | 121.2 (8.2)
Statistical Analysis 1: Comparison: Atenolol vs Nebivolol; Comparing treatment effects on ABPM; Test type: Other — Linear Mixed effect Model, adjusted for baseline values and period effect Difference of LSMeans treatment effect (SE) = -2.59 (1.34); p = 0.06, Linear Mixed effect Model, adjusted for

3. Secondary Outcome: Total Cholesterol
Description: Fasting blood samples were taken at the beginning and end of each treatment period.
Time Frame: Before and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Atenolol | Nebivolol
Number analyzed (Participants) | 44 | 44
mmol/L
  Before | 5.0 (1.0) | 5.1 (0.9)
  After | 4.9 (1.0) | 5.1 (0.9)
Statistical Analysis 1: Comparison: Atenolol vs Nebivolol; Comparing treatment effects on total cholesterol; Test type: Other — Linear Mixed effect Model, adjusted for baseline values and period effect Difference of LSMeans treatment effect (SE) = -0/09 (0.14); p = 0.51, Linear Mixed effect Modelling, adjusted

4. Secondary Outcome: HbA1c
Description: Fasting blood samples were taken at the beginning and end of each treatment period.
Time Frame: Before and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Atenolol | Nebivolol
Number analyzed (Participants) | 44 | 44
percentage of glycosylated hemoglobin
  Before | 5.7 (0.8) | 5.7 (0.8)
  After | 5.7 (0.4) | 5.7 (0.3)
Statistical Analysis 1: Comparison: Atenolol vs Nebivolol; Comparing treatment effects on HbA1c; Test type: Other — Linear Mixed effect Model, adjusted for baseline values and period effect Difference of LSMeans treatment effect (SE) =0.02 (0.03); p = 0.48, Linear Mixed effect Modelling, adjusted

5. Secondary Outcome: BMI
Description: Body weights and heights were taken at the beginning and end of each treatment period.
Time Frame: Before and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Atenolol | Nebivolol
Number analyzed (Participants) | 44 | 44
kg/m^2
  Before | 28.1 (4.6) | 28.2 (4.7)
  After | 28.0 (4.4) | 28.3 (4.7)
Statistical Analysis 1: Comparison: Atenolol vs Nebivolol; Comparing treatment effects on BMI; Test type: Other — Linear Mixed effect Model, adjusted for baseline values and period effect Difference of LSMeans treatment effect (SE) = -0.21(0.13); p = 0.09, Linear Mixed effect Modelling, adjusted

ADVERSE EVENTS:
Time Frame: 32 weeks
Groups:
- Nebivolol 2.5mg Daily: nebivolol 2.5mg daily
  Nebivolol: Nebivolol 25mg daily
Arm/Group | Atenolol 25mg Daily | Nebivolol 2.5mg Daily
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes